CLINICAL TRIAL: NCT02748824
Title: Five-year Incidence of Age-related Macular Degeneration in the Central Region of Portugal
Acronym: AMDIncidencePT
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2016-09; AMDIncidence-CPT (Other: 4C-2016-09)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age- Related Macular Degeneration; Diabetic Retinopathy; Glaucoma; Cataract
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Glaucoma; Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
To assess the five-year incidence of AMD in a population from the central region of Portugal, previously phenotypically characterized.

DETAILED DESCRIPTION:
Subjects who participated in the Epidemiologic Coimbra Eye Study (NCT01298674) between 2009 and 2013 will attend a single visit, after giving informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in the Epidemiologic Coimbra Eye Study (NCT01298674) and that were phenotyped;
* Subjects capable of understanding the information about the study and to give their informed consent to enter the study;
* Subjects willing and able to comply with the study procedures.

Exclusion Criteria:

- Not applicable

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female subjects who have participated and phenotyped in the Epidemiologic Coimbra Eye Study (NTC01298674).
  It is expected to recruit up to a total of 5.996 subjects, that is up to 2.975 subjects from the Mira Healthcare Unit and up to 3.021 subjects from the Lousã Healthcare Unit.
Sampling Method: Non-Probability Sample
Enrollment: 5996 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09-18 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Phenotypic classification of AMD in the five-year clinical visit. Comparison of this classification with the grading of 5 years ago. | 5 years

SECONDARY OUTCOMES:
Risk factors: Demographic, Medical history, Ophthalmologic history, Family history of AMD, Systemic comorbidities and medication, Nutritional and Lifestyle habits. Signs of AMD on the multimodal evaluation. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rufino Silva, PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI/CEC - Centro Ensaios Clínicos, Coimbra, Portugal

REFERENCES:
- [Derived] Barreto P, Farinha C, Coimbra R, Cachulo ML, Melo JB, Lechanteur Y, Hoyng CB, Cunha-Vaz J, Silva R. Interaction between genetics and the adherence to the Mediterranean diet: the risk for age-related macular degeneration. Coimbra Eye Study Report 8. Eye Vis (Lond). 2023 Aug 14;10(1):38. doi: 10.1186/s40662-023-00355-0. PMID 37580831